CLINICAL TRIAL: NCT02779101
Title: Open-label Single Arm Phase II Study on Pembrolizumab for Recurrent Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Study on Pembrolizumab for Recurrent Primary Central Nervous System Lymphoma (PCNSL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Matthias Preusser (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Matthias Preusser, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCNSL01
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Central nervous system lymphoma; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): pembrolizumab
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — Pembrolizumab 200 mg every 3 weeks

SUMMARY:
In summary, there is a high medical need for patients suffering from recurrent/progressive PCNSL. Targeting the PD-1 pathway may represent a very promising novel approach for the treatment of these patients.

DETAILED DESCRIPTION:
The objective of this study are:

PRIMARY OBJECTIVES

* To evaluate the Overall Response Rate (CR/PR) in patients treated with pembrolizumab for relapsed PCNSL after MTX-based first-line therapy
* To evaluate the safety of pembrolizumab in subjects diagnosed with recurrent PCNSL

SECONDARY OBJECTIVES

* To describe Best Overall Response categories (CR, PR, SD, PD) in patients treated with pembrolizumab for relapsed PCNSL after MTX-based first-line therapy
* To describe individual duration of response over time
* To assess progression-free survival in this patient population
* To assess overall survival in this patient population

EXPLORATORY OBJECTIVES

* To assess PD-L1 as a predictive marker for response to pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Minimum of 18 years of age on day of signing informed consent.
* Histologically confirmed diagnosis of PCNSL (DLBCL) at initial diagnosis
* The patient has a Karnofsky performance status of at least 50%.
* Documented progression or recurrence in cranial MRI after prior MTX-based first-line therapy (with or without prior radiotherapy)
* Measurable disease in cranial MRI (lesion size >10x10mm)
* Has no diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment except for a maximum dose of 4 mg/day dexamethasone or equivalent doses of other corticosteroids or control of brain edema, which has been stable or decreased for at least 1 week prior to inclusion.
* Is not pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Female patient of childbearing potential has a negative urine or serum pregnancy test within 24 hours of first pembrolizumab infusion. lf the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* The patient has a life expectancy of at least 3 months.
* The patient has a Karnofsky performance status of at least 50%.
* The patient demonstrates adequate organ function
* Patient is able to undergo Gadolinium-MRI

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Concurrent administration of any other antitumor therapy except steroids
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active infection requiring systemic therapy.
* Known history of active TB (Bacillus Tuberculosis)
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Has received a live vaccine within 30 days of planned start of study therapy.

  o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Drug abuse or extensive use of alcohol.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Positive human immunodeficiency virus (HIV) test and a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* History of allergy to study drug components and no history of severe hypersensitivity reaction to any monoclonal antibody.
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1.
* Has not recovered (i.e.Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Known hypersensitivity to pembrolizumab or any of its excipients.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Response assessment | after 24 month
  Response assessment will be performed according to modified IPCG response criteria on contrast-enhanced cranial MRI-scans

SECONDARY OUTCOMES:
Clinical adverse events | after 24 month
  clinical adverse Events will be assessed by CTCAE v4.0
Laboratory parameters | after 24 month
  adverse events due to laboratory parameters will be assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, MD, Principal Investigator — MU Vienna, Dep. f. Internal medicine I, Oncology
Locations (1):
- Dept of Internal Medicine, Vienna, Austria